CLINICAL TRIAL: NCT00520403
Title: An Open-label Study to Assess the Effect of First-line Treatment With Avastin in Combination With Standard Therapy on Progression-free Survival in Patients With Metastatic Renal Cell Cancer.
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Standard Therapy in Patients With Metastatic Renal Cell Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19983
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Interferon alpha-2; Vinblastine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Interferon alfa-2a; Drug: Vinblastine

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv every 3 weeks
Drug: Interferon alfa-2a — 3 MioIU sc escalating to 18 MioIU sc, 3 times weekly
Drug: Vinblastine — 0.1mg/kg iv every 3 weeks

SUMMARY:
This single arm study will assess the efficacy and safety of Avastin in combination with interferon alfa-2a and vinblastine as first line treatment in patients with metastatic renal cell cancer. Patients will receive Avastin (15mg/kg iv) every 3 weeks, interferon alfa-2a 3 times weekly (3 Mio IU sc escalating to 18 Mio sc) and vinblastine (0.1mg/kg iv) every 3 weeks. The anticipated time on study treatment is until tumor progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* metastatic renal cell cancer of predominantly clear cell type;
* >=1 measurable lesion.

Exclusion Criteria:

* prior treatment with chemotherapy, cytokine or tyrosine kinase inhibitor therapy for metastatic renal cell cancer;
* ongoing or recent need for full therapeutic dose of anticoagulants or chronic daily treatment with aspirin (>325mg/day);
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- Germany (15):
  - Berlin
  - Bremen
  - Dessau
  - Erlangen
  - Frankfurt
  - Halle
  - Hanover
  - Jena
  - Kassel
  - Kiel
  - Leipzig
  - Magdeburg
  - Rehling
  - Stuttgart
  - Weiden

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Interferon Alfa-2a (IFN)/Vinblastine: Cycle 1 (3-week cycle): Participants received vinblastine sulfate 0.1 mg/kg intravenously (IV) and bevacizumab 15 milligrams per kilogram (mg/kg) IV on Day 1 followed by 2 weeks off and IFN subcutaneous (SC) injection three times per week (starting on Day 1) at doses of 3 million International Units (mIU) (Week 1), 9 mIU (Week 2), and 18 mIU (Week 3).
  Cycles 2 to 17 (3-week cycles): Participants received vinblastine sulfate 0.1 mg/kg IV and bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off and IFN 18 mIU SC injection three times per week during Weeks 1 through 3; the cycle was repeated every 3 weeks up to Week 51 (Cycle 17) or to tumor progression.
  If the first 17 cycles were tolerated without tumor progression, participants received bevacizumab monotherapy: bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off; this cycle was repeated every 3 weeks up to Week 102 (Cycle 34) or to tumor progression.
Period: Bevacizumab + IFN/Vinblastine
Arm/Group | Bevacizumab + Interferon Alfa-2a (IFN)/Vinblastine
Started | 25
Completed | 7
Not Completed | 18
Not completed — Radiological progression of cancer | 6
Not completed — Adverse Event | 4
Not completed — Withdrawal of consent | 4
Not completed — Death | 2
Not completed — Discontinuation of study/background drug | 1
Not completed — Protocol Deviation affecting safety | 1
Period: Bevacizumab Monotherapy
Arm/Group | Bevacizumab + Interferon Alfa-2a (IFN)/Vinblastine
Started | 2 (2 of 7 participants completing Bevacizumab+IFN/vinblastine cycles initiated bevacizumab monotherapy)
Completed | 0
Not Completed | 2
Not completed — Radiological progression of cancer | 1
Not completed — Symptomatic progression of cancer | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: included all participants, even those who withdrew from the study prematurely and who received at least 1 dose of bevacizumab and had a safety follow-up visit.
Groups:
- Bevacizumab + IFN/Vinblastine: Cycle 1 (3-week cycle): Participants received vinblastine sulfate 0.1 mg/kg IV and bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off and IFN SC injection three times per week (starting on Day 1) at doses of 3 mIU (Week 1), 9 mIU (Week 2), and 18 mIU (Week 3).
  Cycles 2 to 17 (3-week cycles): Participants received vinblastine sulfate 0.1 mg/kg IV and bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off and IFN 18 mIU SC injection three times per week during Weeks 1 through 3 (starting on Day 1); the cycle was repeated every 3 weeks up to Week 51 (Cycle 17) or to tumor progression.
  If the first 17 cycles were tolerated without tumor progression, participants received bevacizumab monotherapy: bevacizumab 15 mg/kg IV on Day 1 followed by 2 weeks off; this cycle was repeated every 3 weeks up to Week 102 (Cycle 34) or to tumor progression.
Arm/Group | Bevacizumab + IFN/Vinblastine
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression was evaluated according to the Response Evaluation Criteria In Solid Tumors (RECIST) using computed tomography (CT) scans (preferred method), magnetic resonance imaging (MRI) scans, X-ray, bone scans, or clinical examination.
Time Frame: Days 0, 91, 182, 273, 365, 456, and 547
Population: Intent-to-treat (ITT) population: all participants, even those who withdrew from the study prematurely, who received at least 1 dose of study medication and for whom the primary efficacy variable was measured at least once during the time when the participant received study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + IFN/Vinblastine
Number analyzed (Participants) | 17
percentage of participants | 66.9

2. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based on assessment of confirmed complete remission (CR) or confirmed partial remission (PR) according to RECIST.
Time Frame: Baseline and Cycles 3, 6, 9, 13, and 17
Population: ITT Population; missing data were imputed using the last observation carried forward (LOCF) technique. Number (n) equals (=) number of participants assessed at each specific visit.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + IFN/Vinblastine
Number analyzed (Participants) | 17
percentage of participants
  Week 9 (n=14) | 21.4
  Week 18 (n=16) | 31.3
  Week 27 (n=16) | 37.5
  Week 39 (n=16) | 31.3
  Week 51 (n=16) | 31.3

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from treatment start to death from any cause. Overall survival was censored at the last contact for surviving participants and missing data points.
Time Frame: Baseline, Day 1 of every cycle to disease progression or death (up to Week 102)
Population: Two of 25 participants died during the course of the study, thus, median overall survival could not be analyzed.
Measure: Median (Full Range); unit: weeks
Arm/Group | Bevacizumab + IFN/Vinblastine
Number analyzed (Participants) | 25
weeks | NA [NA to NA] — Median could not be calculated due to lack of events as only 2 of 25 participants died during the course of the study.

4. Primary Outcome: PFS - Time to Event
Description: PFS was defined as the time in days from the date of treatment start to the date of first documented disease progression or death. Disease progression was evaluated according to RECIST using CT scans (preferred method), MRI scans, X-ray, bone scans, or clinical examination. Median PFS was estimated using the Kaplan-Meier method
Time Frame: Days 0, 91, 182, 273, 365, 456, and 547
Population: ITT population.
Measure: Median (Standard Error); unit: days
Arm/Group | Bevacizumab + IFN/Vinblastine
Number analyzed (Participants) | 17
days | 274 (31.6)

ADVERSE EVENTS:
Time Frame: From treatment start to 28 days after treatment cessation in the regular treatment period only (Cycles 1 through 17; bevacizumab + IFN/vinblastine). Does not include AEs reported during bevacizumab monotherapy (Cycles 18 and beyond).
Description: AE (serious and non-serious) information was collected for participants in the Safety Population and reported for the regular treatment period only (Cycles 1 through 17; bevacizumab + IFN/vinblastine).
Arm/Group | Bevacizumab + IFN/Vinblastine
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + IFN/Vinblastine (N=25)
Neutropenia (Blood and lymphatic system disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
General Physical Health Deterioration (General disorders) | 1
Injection Site Reaction (General disorders) | 1
Systemic Inflammatory Response Syndrome (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + IFN/Vinblastine (N=25)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Ileus paralytic (Gastrointestinal disorders) | 1
Loose tooth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Periodontitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Tongue ulceration (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 5
Drug intolerance (General disorders) | 1
Fatigue (General disorders) | 10
Impaired healing (General disorders) | 1
Influenza like illness (General disorders) | 6
Mucosal inflammation (General disorders) | 4
Pyrexia (General disorders) | 3
Abscess jaw (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood sodium decreased (Investigations) | 1
Intraocular pressure test (Investigations) | 1
Urine output decreased (Investigations) | 1
Weight decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Fascial hernia (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depressed mood (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 8
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Scar pain (Skin and subcutaneous tissue disorders) | 2
Skin atrophy (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.